CLINICAL TRIAL: NCT04319029
Title: Assessment of Patients' Knowledge, Quality of Life, and Adherence for Medication in Dyslipidemia - a Randomized Interventional Study
Brief Title: Assessment of Dyslipidemic Patients' Knowledge, Quality of Life, and Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AR190101
Record Dates: First submitted 2020-03-13; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-intervention (No Intervention): Patients received a conventional pharmaceutical care plan, the patients offered optimal pharmacological therapy wit statin.
- Intervention (Active Comparator): The Patients offered to predesign pharmaceutical care plans aimed to improved patient's knowledge, adherence, satisfaction, and quality of life. The patients offered optimal pharmacological therapy wit statin.
  Interventions: Behavioral: Pharmaceutical care plan

INTERVENTIONS:
Behavioral: Pharmaceutical care plan — The design of the intervention was based on a stepwise approach to address the following point in each participant: set priorities for patient care, assessment of patient's educational needs, and development of a comprehensive and achievable pharmaceutical care plan.
  The participants will be educated about their illness and informed about the proper use of their medication in a structured manner (it involved the following items: dyslipidemia as a disease, complications, who therapy reduces its risk and complications, goal of therapy). Behavioral modifications will involve the following: physical exercise, diet, smoking cessation. Patients will obtain this information verbally and provided in a written manner through a brochure that design for this study.
  Arms: Intervention

SUMMARY:
A randomized, parallel two-arm interventional study, the patients were divided into 1:1 ratio, in which both groups offered optimal pharmacological therapy also one group (interventional) offered predesign pharmaceutical care plan aimed to improved patients knowledge, adherence, satisfaction, and quality of life, while the other group (non-interventional) received conventional pharmaceutical care plan.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with dyslipidemia and received at least one statin therapy (in the previous 6 months), and patients on the same class of pharmacological therapy (statins).

Exclusion Criteria:

1. Pregnant women
2. Nephrotic syndrome
3. Active steroid user
4. Hypersensitivity for any mediation during the trial
5. History of a major cardiovascular event in the previous 3 months
6. Patients with mental disease or disability
7. Had a stroke in the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the patient satisfaction | Baseline, and At 6 months
  Pharmaceutical Care Satisfaction Questionnaire (PCSQ) score for patient satisfaction:
  A 30-items score each item composed of a 5-point Likert scale (5 = strongly agree and 1 = strongly disagree), then the items are averaged and presented (value between 1 - 5) Unit of Measure is units on a Scale of 5
Change in the medication adherence in intervention group vs. non-intervention group | Baseline, at 3 months, and at 6 months
  Visual Analogue Scale (VAS) for medication adherence:
  The participants will be asked to mark a line at the point along a continuum showing how much of each drug they have taken in the past month, this scare take range from 0 - 10.
  Unit of Measure is units on a Scale of 10
Change in the hyperlipidemia-Patient Knowledge in intervention group vs. non-intervention group | Baseline, and At 6 months
  Hyperlipidemia-Patient Knowledge Evaluation score:
  The Hyperlipidemia-Patient Knowledge Evaluation is a 17-item true-or-false questionnaire, which involved general knowledge, habit, diet, pharmacotherapy, and complications. The score ranges from 0 - 16.
  Unit of Measure is units on a Scale of 16
Change in the quality of life in intervention group vs. non-intervention group | Baseline, and At 6 months
  The RAND 36-items score (SF-36) for quality of life (QoL):
  This score composed of 36-items that contain 8 domains, the score has a range from 0 - 100 which represents the average of these domains.
  Unit of Measure is units on a Scale of 100

SECONDARY OUTCOMES:
Change in Serum LDL in intervention group vs. non-intervention group | Baseline, and At 6 months
  Change in serum LDL that will occur in both the intervention group and non-intervention group, and determine which group will provide a more significant reduction in serum LDL.
  Unit of Measure is mg/dL
Change in Serum HDL in intervention group vs. non-intervention group | Baseline, and At 6 months
  Change in serum HDL that will occur in both the intervention group and non-intervention group, and determine which group will provide a more significant reduction in serum HDL.
  Unit of Measure is mg/dL
Change in Serum cholesterol in intervention group vs. non-intervention group | Baseline, and At 6 months
  Change in serum cholesterol that will occur in both the intervention group and non-intervention group, and determine which group will provide a more significant reduction in serum HDL.
  Unit of Measure is mg/dL
Rate of Medication-related problems manged | Up to 6 months
  Each successful management of medication-related problems reported by the patients by the pharmacist will be recorded and compared between the intervention group vs. non-intervention group Unit of measure is the percentage

CONTACTS AND LOCATIONS:
Overall Officials: Hayder F Al-Tukmagi, PhD, Principal Investigator — Al-Mustaffa University College; Hayder A Fawzi, PhD, Study Chair — Al-Rasheed University College
Locations (1):
- Al-Rasheed University College, Baghdad, AL-Adhmia, Iraq

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Starting after the publication of the research
Access Criteria: Any interested Party